CLINICAL TRIAL: NCT06166641
Title: Prediction Models for Risk Score and Prognosis of Intraoperatively Acquired Pressure Injury in Surgical Patients: a Multicenter Prospective Cohort Study
Brief Title: Prediction Models for Risk Score and Prognosis of Intraoperatively Acquired Pressure Injury in Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Guangdong Medical University (Other)
Responsible Party: Principal Investigator, Yiyue Zhong, Nursing Supervisory, Affiliated Hospital of Guangdong Medical University
Other Study IDs: PJKT2023-007
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-06

CONDITIONS: Pressure Ulcer; Predictive Models; Surgical Patient; Clinical Outcome
Keywords: intraoperatively acquired pressure injury; Pressure Ulcer; predictive models; surgical patient; clinical outcome
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intraoperative acquired pressure injury: Intraoperative acquired pressure injury are wounds that develop during a surgical procedure or while a patient is in the operating room. These ulcers are caused by prolonged pressure on a specific area of the body, which reduces blood flow and leads to tissue damage.
  Interventions: Procedure: Surgical procedure at operating room

INTERVENTIONS:
Procedure: Surgical procedure at operating room — A surgical procedure in an operating room is a medical intervention that involves making incisions or using minimally invasive techniques to treat a specific condition or perform a diagnostic procedure. The operating room, also known as the operating theater or surgical suite, is a sterile environment specifically designed to minimize the risk of infection and ensure the safety of both the patient and the surgical team.

SUMMARY:
The study aims to effectively identify the risk of intraoperative acquired pressure injuries (IAPI) in surgical patients through a prospective multicenter approach. It combines indicators from commonly used assessment tools and practical experience judgments to construct a comprehensive assessment framework.

By incorporating various indicators, the study aims to improve the accuracy and reliability of identifying patients at risk of IAPI during surgery. This will help clinicians in making informed decisions and implementing preventive measures to minimize the occurrence of pressure injuries.

The multicenter approach ensures a diverse and representative sample of patients from different surgical settings. This increases the generalizability of the study findings and enhances the applicability of the assessment framework across various clinical settings.

The project's methodology involves collecting data on patient demographics, medical history, surgical procedure details, and assessment tool scores. These data points will be analyzed to identify significant risk factors for IAPI and develop a risk prediction model.

The study also takes into consideration practical experience judgments, which acknowledge the importance of clinical expertise in assessing patients' risk of IAPI. This ensures that the assessment framework is not solely reliant on assessment tools but also incorporates the insights of experienced clinicians.

Overall, this prospective multicenter study aims to contribute to the field by providing a comprehensive and practical approach to identify the risk of IAPI in surgical patients. The findings from this study can be utilized in clinical practice to improve patient outcomes and reduce the incidence of pressure injuries during surgery.

ELIGIBILITY:
Inclusion criteria: All patients who underwent surgery procedure at the participating setting after the study registration.

Exclusion criteria: Patients who have already been diagnosed with pressure injury (stage II and above) before undergoing surgery procedure. Patients/relatives/guardians understand the refusal of data to be used for clinically relevant research. Investigators believe that certain patient conditions may affect the efficacy and safety assessment of this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The inclusion and exclusion criteria provided suggest that the study aims to evaluate the clinical characteristic of pressure injury in patients who undergo surgery. The study will include all patients who undergo surgery at the participating setting after study registration. This broad inclusion criteria allows for a diverse patient population to be included in the study.
Sampling Method: Probability Sample
Enrollment: 5658 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative acquired pressure injury | Perioperative Period
  Intraoperative acquired pressure injuries, also known as intraoperative pressure ulcers or surgical pressure injuries, are wounds that develop during a surgical procedure. These injuries occur due to prolonged pressure on specific areas of the body, which disrupts blood flow and leads to tissue damage.

SECONDARY OUTCOMES:
Mortality | Perioperative Period
  All deaths reported in the study population

CONTACTS AND LOCATIONS:
Overall Officials: Yiyue Zhong, MD, Principal Investigator — Affiliated Hospital of Guangdong Medical University
Locations (1):
- The Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
The data sharing policies and decisions are typically determined by the researchers or organizations conducting the study, in collaboration with any relevant ethical review boards and regulatory bodies.

REFERENCES:
- [Result] Dunk AM, Carville K. The international clinical practice guideline for prevention and treatment of pressure ulcers/injuries. J Adv Nurs. 2016 Feb;72(2):243-4. doi: 10.1111/jan.12614. Epub 2015 Jan 6. No abstract available. PMID 25558893
- [Result] Xiong C, Gao X, Ma Q, Yang Y, Wang Z, Yu W, Yu L. Risk factors for intraoperative pressure injuries in patients undergoing digestive surgery: A retrospective study. J Clin Nurs. 2019 Apr;28(7-8):1148-1155. doi: 10.1111/jocn.14712. Epub 2018 Dec 7. PMID 30375697
- [Result] Nixon J, Brown J, McElvenny D, Mason S, Bond S. Prognostic factors associated with pressure sore development in the immediate post-operative period. Int J Nurs Stud. 2000 Aug;37(4):279-89. doi: 10.1016/s0020-7489(99)00059-0. PMID 10760535
- [Result] Gillespie BM, Walker RM, Latimer SL, Thalib L, Whitty JA, McInnes E, Lockwood I, Chaboyer WP. Repositioning for pressure injury prevention in adults: An abridged Cochrane systematic review and meta-analysis. Int J Nurs Stud. 2021 Aug;120:103976. doi: 10.1016/j.ijnurstu.2021.103976. Epub 2021 May 18. PMID 34090235
- [Result] Gillespie BM, Walker RM, Latimer SL, Thalib L, Whitty JA, McInnes E, Chaboyer WP. Repositioning for pressure injury prevention in adults. Cochrane Database Syst Rev. 2020 Jun 2;6(6):CD009958. doi: 10.1002/14651858.CD009958.pub3. PMID 32484259
- [Result] Gallagher P, Barry P, Hartigan I, McCluskey P, O'Connor K, O'Connor M. Prevalence of pressure ulcers in three university teaching hospitals in Ireland. J Tissue Viability. 2008 Nov;17(4):103-9. doi: 10.1016/j.jtv.2007.12.001. Epub 2008 Apr 18. PMID 18378140
- [Result] Vazykhova FG, Viazov SO, Anan'ev VA. [Polypeptide composition of the delta-antigen]. Vopr Virusol. 1989 May-Jun;34(3):299-302. Russian. PMID 2477952
- [Result] Labeau SO, Afonso E, Benbenishty J, Blackwood B, Boulanger C, Brett SJ, Calvino-Gunther S, Chaboyer W, Coyer F, Deschepper M, Francois G, Honore PM, Jankovic R, Khanna AK, Llaurado-Serra M, Lin F, Rose L, Rubulotta F, Saager L, Williams G, Blot SI; DecubICUs Study Team; European Society of Intensive Care Medicine (ESICM) Trials Group Collaborators. Correction to: Prevalence, associated factors and outcomes of pressure injuries in adult intensive care unit patients: the DecubICUs study. Intensive Care Med. 2021 Apr;47(4):503-520. doi: 10.1007/s00134-020-06327-5. No abstract available. PMID 33635356
- [Result] Nguyen HL, Vu VC, Nguyen DL, Vo HL, Nguyen QD. Posterior surgical approach for the treatment of lower cervical spine injury with spinal cord paralysis: high postoperative mortality in resource-scare setting. Eur Rev Med Pharmacol Sci. 2022 Apr;26(8):2960-2969. doi: 10.26355/eurrev_202204_28627. PMID 35503640
- [Result] Hopkins A, Dealey C, Bale S, Defloor T, Worboys F. Patient stories of living with a pressure ulcer. J Adv Nurs. 2006 Nov;56(4):345-53. doi: 10.1111/j.1365-2648.2006.04007.x. PMID 17042814
- [Result] Khor HM, Tan J, Saedon NI, Kamaruzzaman SB, Chin AV, Poi PJ, Tan MP. Determinants of mortality among older adults with pressure ulcers. Arch Gerontol Geriatr. 2014 Nov-Dec;59(3):536-41. doi: 10.1016/j.archger.2014.07.011. Epub 2014 Jul 21. PMID 25091603
- [Result] Manzano F, Perez-Perez AM, Martinez-Ruiz S, Garrido-Colmenero C, Roldan D, Jimenez-Quintana Mdel M, Sanchez-Cantalejo E, Colmenero M. Hospital-acquired pressure ulcers and risk of hospital mortality in intensive care patients on mechanical ventilation. J Eval Clin Pract. 2014 Aug;20(4):362-8. doi: 10.1111/jep.12137. Epub 2014 May 22. PMID 24854297
- [Result] Bauer K, Rock K, Nazzal M, Jones O, Qu W. Pressure Ulcers in the United States' Inpatient Population From 2008 to 2012: Results of a Retrospective Nationwide Study. Ostomy Wound Manage. 2016 Nov;62(11):30-38. PMID 27861135
- [Result] EXTON-SMITH AN, SHERWIN RW. The prevention of pressure sores. Significance of spontaneous bodily movements. Lancet. 1961 Nov 18;2(7212):1124-6. doi: 10.1016/s0140-6736(61)91033-9. No abstract available. PMID 13891095
- [Result] Waterlow J. Pressure sores: a risk assessment card. Nurs Times. 1985 Nov 27-Dec 3;81(48):49-55. No abstract available. PMID 3853163
- [Result] Waterlow J. Tissue viability. Prevention is cheaper than cure. Nurs Times. 1988 Jun 22-28;84(25):69-70. No abstract available. PMID 3405804
- [Result] Waterlow J. A policy that protects. The Waterlow Pressure Sore Prevention/Treatment Policy. Prof Nurse. 1991 Feb;6(5):258, 260, 262-4. PMID 2000416
- [Result] Braden B, Bergstrom N. A conceptual schema for the study of the etiology of pressure sores. Rehabil Nurs. 1987 Jan-Feb;12(1):8-12. doi: 10.1002/j.2048-7940.1987.tb00541.x. No abstract available. PMID 3643620
- [Result] Hunt J. Application of a pressure area risk calculator in an intensive care unit. Intensive Crit Care Nurs. 1993 Dec;9(4):226-31. doi: 10.1016/s0964-3397(05)80003-5. PMID 8274831
- [Result] Qaseem A, Mir TP, Starkey M, Denberg TD; Clinical Guidelines Committee of the American College of Physicians. Risk assessment and prevention of pressure ulcers: a clinical practice guideline from the American College of Physicians. Ann Intern Med. 2015 Mar 3;162(5):359-69. doi: 10.7326/M14-1567. PMID 25732278
- [Result] Munro CA. The development of a pressure ulcer risk-assessment scale for perioperative patients. AORN J. 2010 Sep;92(3):272-87. doi: 10.1016/j.aorn.2009.09.035. PMID 20816101
- [Result] Wang LH, Chen HL, Yan HY, Gao JH, Wang F, Ming Y, Lu L, Ding JJ. Inter-rater reliability of three most commonly used pressure ulcer risk assessment scales in clinical practice. Int Wound J. 2015 Oct;12(5):590-4. doi: 10.1111/iwj.12376. Epub 2014 Sep 16. PMID 25224688
- [Result] Anthony D, Parboteeah S, Saleh M, Papanikolaou P. Norton, Waterlow and Braden scores: a review of the literature and a comparison between the scores and clinical judgement. J Clin Nurs. 2008 Mar;17(5):646-53. doi: 10.1111/j.1365-2702.2007.02029.x. PMID 18279297
- [Result] Schoonhoven L, Haalboom JR, Bousema MT, Algra A, Grobbee DE, Grypdonck MH, Buskens E; prePURSE study group. The prevention and pressure ulcer risk score evaluation study. Prospective cohort study of routine use of risk assessment scales for prediction of pressure ulcers. BMJ. 2002 Oct 12;325(7368):797. doi: 10.1136/bmj.325.7368.797. PMID 12376437
- [Result] Moore ZE, Patton D. Risk assessment tools for the prevention of pressure ulcers. Cochrane Database Syst Rev. 2019 Jan 31;1(1):CD006471. doi: 10.1002/14651858.CD006471.pub4. PMID 30702158
- [Result] Jun Seongsook RN, Jeong Ihnsook RN, Lee Younghee RN. Validity of pressure ulcer risk assessment scales; Cubbin and Jackson, Braden, and Douglas scale. Int J Nurs Stud. 2004 Feb;41(2):199-204. doi: 10.1016/s0020-7489(03)00135-4. PMID 14725784
- [Result] Higgins J, Casey S, Taylor E, Wilson R, Halcomb P. Comparing the Braden and Jackson/Cubbin Pressure Injury Risk Scales in Trauma-Surgery ICU Patients. Crit Care Nurse. 2020 Dec 1;40(6):52-61. doi: 10.4037/ccn2020874. PMID 33257967
- [Result] Gul A, Sengul T, Yavuz HO. Assessment of the risk of pressure ulcer during the perioperative period: Adaptation of the Munro scale to Turkish. J Tissue Viability. 2021 Nov;30(4):559-565. doi: 10.1016/j.jtv.2021.06.009. Epub 2021 Jul 1. PMID 34312031
- [Result] Lei L, Zhou T, Xu X, Wang L. Munro Pressure Ulcer Risk Assessment Scale in Adult Patients Undergoing General Anesthesia in the Operating Room. J Healthc Eng. 2022 Mar 21;2022:4157803. doi: 10.1155/2022/4157803. eCollection 2022. PMID 35356613
- [Result] Bruno R, Bertolino D, Garbarino E, Munro CA, Barisone M, Dal Molin A. Translation, cross-cultural adaptation, and validation of the Munro Scale in Italian. Wound Manag Prev. 2022 Feb;68(2):34-41. PMID 35343919
- [Result] Goras C, Unbeck M, Nilsson U, Ehrenberg A. Interprofessional team assessments of the patient safety climate in Swedish operating rooms: a cross-sectional survey. BMJ Open. 2017 Sep 1;7(9):e015607. doi: 10.1136/bmjopen-2016-015607. PMID 28864690
- [Result] Berrios-Torres SI, Umscheid CA, Bratzler DW, Leas B, Stone EC, Kelz RR, Reinke CE, Morgan S, Solomkin JS, Mazuski JE, Dellinger EP, Itani KMF, Berbari EF, Segreti J, Parvizi J, Blanchard J, Allen G, Kluytmans JAJW, Donlan R, Schecter WP; Healthcare Infection Control Practices Advisory Committee. Centers for Disease Control and Prevention Guideline for the Prevention of Surgical Site Infection, 2017. JAMA Surg. 2017 Aug 1;152(8):784-791. doi: 10.1001/jamasurg.2017.0904. PMID 28467526
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Timsit JF, Ruppe E, Barbier F, Tabah A, Bassetti M. Bloodstream infections in critically ill patients: an expert statement. Intensive Care Med. 2020 Feb;46(2):266-284. doi: 10.1007/s00134-020-05950-6. Epub 2020 Feb 11. PMID 32047941
- [Result] Riley RD, Ensor J, Snell KIE, Harrell FE Jr, Martin GP, Reitsma JB, Moons KGM, Collins G, van Smeden M. Calculating the sample size required for developing a clinical prediction model. BMJ. 2020 Mar 18;368:m441. doi: 10.1136/bmj.m441. No abstract available. PMID 32188600
- [Result] Riley RD. Correction to: Minimum sample size for developing a multivariable prediction model: Part II-binary and time-to-event outcomes by Riley RD, Snell KI, Ensor J, et al. Stat Med. 2019 Dec 30;38(30):5672. doi: 10.1002/sim.8409. Epub 2019 Oct 29. No abstract available. PMID 31793031
- [Result] Guo Y, Zhao K, Zhao T, Li Y, Yu Y, Kuang W. The effectiveness of curvilinear supine position on the incidence of pressure injuries and interface pressure among surgical patients. J Tissue Viability. 2019 May;28(2):81-86. doi: 10.1016/j.jtv.2019.02.005. Epub 2019 Feb 25. PMID 30878174
- [Result] Porter-Armstrong AP, Moore ZE, Bradbury I, McDonough S. Education of healthcare professionals for preventing pressure ulcers. Cochrane Database Syst Rev. 2018 May 25;5(5):CD011620. doi: 10.1002/14651858.CD011620.pub2. PMID 29800486
- [Result] Leary M, Villarruel AM, Richmond TS. Creating an innovation infrastructure in academic nursing. J Prof Nurs. 2022 Jan-Feb;38:83-88. doi: 10.1016/j.profnurs.2021.12.005. Epub 2021 Dec 16. PMID 35042594
- [Result] Rosen J, Mittal V, Degenholtz H, Castle N, Mulsant BH, Hulland S, Nace D, Rubin F. Ability, incentives, and management feedback: organizational change to reduce pressure ulcers in a nursing home. J Am Med Dir Assoc. 2006 Mar;7(3):141-6. doi: 10.1016/j.jamda.2005.08.003. Epub 2005 Dec 12. PMID 16503306
- [Result] Stulberg JJ, Huang R, Kreutzer L, Ban K, Champagne BJ, Steele SR, Johnson JK, Holl JL, Greenberg CC, Bilimoria KY. Association Between Surgeon Technical Skills and Patient Outcomes. JAMA Surg. 2020 Oct 1;155(10):960-968. doi: 10.1001/jamasurg.2020.3007. PMID 32838425

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT06166641/Prot_SAP_000.pdf